CLINICAL TRIAL: NCT00769769
Title: Telephone CBT for Depressed African-American Dementia Caregivers
Brief Title: Comparing Delivery Methods of Cognitive Behavioral Therapy for Depressed African-American Dementia Caregivers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Robert L. Glueckauf (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Robert L. Glueckauf, Principal Investigator, Florida State University
Organization: Florida State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH078999 (NIH); R34MH078999 (NIH); DATR A4-GPS
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Depression
Keywords: Health Status
MeSH Terms: conditions — Depression | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone-based psychotherapy (Experimental)
  Interventions: Behavioral: Psychotherapy
- Face-to-face psychotherapy (Active Comparator)
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Participants will receive 12 sessions of cognitive behavioral therapy delivered weekly over a period of 3 months.
  Arms: Face-to-face psychotherapy
Behavioral: Psychotherapy — Participants will receive 12 sessions of telephone-based cognitive behavioral therapy delivered weekly over 3 months.
  Arms: Telephone-based psychotherapy

SUMMARY:
This study will compare the effectiveness of face-to-face cognitive behavioral therapy versus telephone-based cognitive behavioral therapy for treating African Americans who care for family members with dementia.

DETAILED DESCRIPTION:
Approximately 4.5 million Americans suffer from progressive dementia, with higher rates among African Americans than among European Americans. The majority of caregivers for dementia patients are family members, who often deal with difficult behavior, agitation, and aggressiveness in the people for whom they care. Because of the challenges they face, family caregivers for dementia patients are at increased risk of mental health problems, particularly depression. Promising research has shown that cognitive behavioral therapy (CBT) can combat distress in African-American caregivers. One way to deliver CBT is through telephone-based interventions, which have been shown to lead to better psychological outcomes than routine education and support. This study will create treatment manuals for CBT tailored to the needs and preferences of African Americans who care for family members with dementia and will develop procedures and strategies for treatment delivery to and retention of members of this population. The study will then compare the effectiveness of face-to-face versus telephone-based CBT in improving mental health outcomes for African Americans who care for family members with dementia.

Participation in this study will last 3 months. Participants will be randomly assigned to receive either face-to-face or telephone-based CBT. Both groups will receive 12 weekly sessions of therapy targeting caregiver depression and social functioning over time. Before and after treatment, participants will be assessed on measures of depression and social functioning through standardized questionnaires given over the telephone. Additional data will be collected on social and demographic factors, stressors, caregiver appraisal of resources, and use and costs of both mental and physical health care.

ELIGIBILITY:
Inclusion Criteria:

* Provides significant care for a spouse, parent, or relative who meets National Institute of Neurological and Communicative Disorders and Strokes-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for probable dementia
* Provides care for a relative 60 years of age or older with progressive dementia
* Primary informal care provider for the care recipient with dementia
* Spends a minimum of 6 hours per week in providing direct care to the person with progressive dementia
* Scores a minimum of 10 on the Patient Health Questionnaire-9 (PHQ-9)

Exclusion Criteria:

* Endorses fewer than three problems on the depression and disruptive behaviors factors of the modified version of Revised Memory and Behavior Problem Checklist
* Meets criteria for psychotic disorder on the Mini-International Neuropsychiatric Interview (MINI 5.0.0)
* Meets criteria for moderate or high suicide risk on the MINI 5.0.0
* Provides care for a dementia care recipient who has received a terminal diagnosis of 6 months, as defined by hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Depression clinical diagnosis | Measured before and after 3-month intervention

SECONDARY OUTCOMES:
Caregiver health status | Measured before and after 3-month intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Glueckauf, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University College of Medicine, Tallahassee, Florida, United States